CLINICAL TRIAL: NCT05633459
Title: A Multi-Center, Randomized, Double-Blind Placebo Controlled Multiple-Ascending Dose Study to Evaluate the Safety and Tolerability of QRL-201 in Amyotrophic Lateral Sclerosis
Brief Title: A Study Evaluating the Safety and Tolerability of QRL-201 in ALS
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: QurAlis Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QRL-201-01
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS, Stathmin-2, STMN2, ASO, Antisense Oligonucleotide
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Masking Description: Multiple-ascending doses of QRL-201 or placebo will be administered. The dose levels may change subject to available nonclinical, clinical, safety, and PK data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- QRL-201: Sporadic ALS (Experimental): Multiple-ascending doses of QRL-201 will be intrathecally administered to individuals with ALS.
  Interventions: Drug: Multiple ascending doses of QRL-201
- Placebo: Sporadic ALS (Placebo Comparator): Multiple-ascending doses of placebo comparator will be intrathecally administered to individuals with ALS.
  Interventions: Drug: Multiple ascending doses of Placebo
- QRL-201: C9orf72-ALS (Experimental): QRL-201 will be intrathecally administered to individuals with C9orf72-ALS.
  Interventions: Drug: QRL-201
- Placebo: C9orf72-ALS (Placebo Comparator): Placebo comparator will be intrathecally administered to individuals with C9orf72-ALS.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Multiple ascending doses of QRL-201 — Multiple ascending doses of QRL-201 will be intrathecally administered to individuals with sporadic ALS.
  Arms: QRL-201: Sporadic ALS
Drug: Multiple ascending doses of Placebo — Multiple ascending doses of placebo comparator will be intrathecally administered to individuals with sporadic ALS.
  Arms: Placebo: Sporadic ALS
Drug: QRL-201 — QRL-201 will be intrathecally administered to individuals with C9orf72 ALS.
  Arms: QRL-201: C9orf72-ALS
Drug: Placebo — Placebo comparator will be intrathecally administered to individuals with C9orf72 ALS.
  Arms: Placebo: C9orf72-ALS

SUMMARY:
The primary objective of this study is to determine the safety and tolerability of multiple doses of QRL-201 in people living with ALS

DETAILED DESCRIPTION:
This first-in-human, Phase 1 study will evaluate the safety, tolerability, and pharmacokinetics (PK) of QRL-201 administered intrathecal (IT) to participants with Amyotrophic Lateral Sclerosis. Two dose escalation cohorts of 8 participants each, followed by an additional 48 participants, receiving the study drug in a 6:2 ratio of QRL-201 to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 18 to 80 years diagnosed with ALS
* ALS symptom onset within 24 months of Screening
* Slow vital capacity >50%
* Clinical or electrodiagnostic evidence of lower motor neuron involvement
* Not pregnant and not nursing
* Willing and able to practice effective contraception
* Able to tolerate lumbar puncture
* If on approved therapies for the treatment of ALS during the course of the study, must be on a stable dose (at the Sponsor's discretion)

Exclusion Criteria:

* Pathogenic variant, likely pathogenic variant, or variant of uncertain significance in the superoxide dismutase 1 (SOD1) and/or fused in sarcoma (FUS) genes
* Currently enrolled in any other clinical study involving either an investigational product (IP) or off-label use of a drug or device
* Prior exposure to stem cell or gene therapy products
* Any contraindication to intrathecal drug administration
* Abnormal laboratory values deemed clinically significant by the Investigator
* Significant infection or known inflammatory process
* Any sign and/or history of neurological conditions and other neuromuscular disorders that could affect the electrophysiological recordings.
* An EEG that shows signs of abnormal electrical activity (e.g., epilepsy)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-12-16 (Actual); Primary Completion 2026-10-08 (Estimated); Study Completion 2026-10-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with one or more treatment emergent adverse events and serious adverse events | Baseline through Day 421 [End of Study Visit
  Endpoints: A summary of treatment emergent adverse events, serious adverse events, and other non-serious adverse events, regardless of causality, will be reported in the Reported Adverse Events module.

SECONDARY OUTCOMES:
Pharmacokinetics (plasma): Maximum observed concentration of QRL-201 (Cmax) | Predose up to 24 hours post dose
  Endpoints: PK: Cmax of QRL-201
Pharmacokinetics (plasma): Area under the concentration time curve from zero to infinity (AUCinf) of QRL-201 | Predose up to 24 hours post dose
  Endpoints: PK: AUC (0-inf) of QRL-201
Pharmacokinetics (plasma): Time of maximum concentration (Tmax) of QRL-201 | Predose up to 24 hours postdose
  Endpoints: PK: Tmax of QRL-201

CONTACTS AND LOCATIONS:
Overall Officials: Angela Genge, MD, Study Director — QurAlis Corporation
Locations (15):
- Universitaire Ziekenhuizen Leuven (UZ Leuven), Leuven, Belgium
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - Montreal Neurological Institute-Hospital, Montreal, Quebec
- Germany (4):
  - Deutsches Zentrum für Neurodegenerative Erkrankungen e. V. (DZNE), Bonn, North Rhine-Westphalia
  - Charité Research Organisation, Berlin
  - University Hospital Schleswig-Holstein (UKSH) Campus Lübeck, Department for Neurology/ Precision Neurology, Lübeck
  - Universitätsklinikum Ulm, Ulm
- St James's Hospital, Dublin, Ireland
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- United Kingdom (3):
  - The University of Sheffield, Royal Hallamshire Hospital, Sheffield, United Kingdom
  - Kings College Hospital NHS Foundation Trust, London
  - National Hospital for Neurology and Neurosurgery, London

IPD SHARING:
Plan to Share IPD: No